CLINICAL TRIAL: NCT06774547
Title: The Efficacy of Early Implementation of Plyometric Exercises in the Rehabilitation of Individuals Suffering From Lower-Extremity Tendinopathies: A Randomised Clinical Trial
Brief Title: Early Implementation of Plyometric Exercises in the Rehabilitation of Individuals Suffering From Lower-Extremity Tendinopathies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Department of Physiotherapy, University College of Northern Denmark (Unknown)
Responsible Party: Principal Investigator, Henrik Riel, Postdoc, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20240042
Record Dates: First submitted 2025-01-03; First posted 2025-01-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Achilles Tendinopathy; Patellar Tendinopathy; Plantar Fasciopathy
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometrics (Experimental): Performing both heavy-slow resistance training and the plyometric protocol
  Interventions: Other: Heavy-slow resistance training; Other: Plyometric exercise
- Control (Active Comparator): Perform heavy-slow resistance training
  Interventions: Other: Heavy-slow resistance training

INTERVENTIONS:
Other: Heavy-slow resistance training — Heavy-slow resistance training consists of a progressive protocol of dynamic exercises where the relative load increases over time from a weight that can only be lifted 15 times (i.e., 15 repetition maximum) during the first week to a relative load of 6 repetition maximum from Week 9 to 12. The exercises are performed unsupervised three days per week separated by a minimum of 48 hours. There are two exercises that are performed for four sets separated by a 2-minute rest. Participants with Achilles tendinopathy or plantar fasciopathy perform seated and standing weighted heel raises and participants with patellar tendinopathy perform a free-standing squat and a seated leg press. Tolerable pain during the exercises is allowed.
Other: Plyometric exercise — The progressive plyometric programme consists of three different levels and is performed unsupervised three times per week separated by a minimum of 48 hours. Each level consists of several exercise sets that are separated by 2-minute rest intervals. Participants' self-evaluated readiness to progress to a higher level will guide the progression. Level 1 includes free-standing double-legged plyometric exercises where they push off the ground and lift their heels while maintaining contact with it. If the participant feels they can do more, they will progress to Level 2, where participants increase the relative load during the dynamic exercises and start performing plyometric double-legged jumps. At the highest level, Level 3, the relative load during the exercises is further increased, and the plyometric exercises are to be performed as single-legged hops. Tolerable pain during the exercises is allowed.
  Arms: Plyometrics

SUMMARY:
This clinical trial aims to compare the effectiveness of an early plyometric exercise approach with traditional heavy, slow resistance training in treating tendinopathies of the Achilles tendon, patellar tendon, and plantar fascia. These conditions, commonly seen in general and rheumatology practices, cause pain, reduced function, and stiffness, often leading to prolonged recovery and incomplete return to full physical activity. The study hypothesizes that introducing plyometric exercises early in rehabilitation will improve jump function after 12 weeks and reduce re-injury rates within 52 weeks compared to traditional methods.

The study is a randomized clinical trial including 120 participants aged 18-50 with tendinopathy in one of the targeted areas. Participants must regularly engage in running or jumping sports, have symptoms for at least three months, and meet other inclusion criteria. Exclusion criteria include recent surgery or specific medical conditions. Both groups will perform exercises three times weekly for 12 weeks, tailored to their tendinopathy. The intervention group will add progressive plyometric exercises to the standard strength training performed by the control group. Plyometric training will consist of three levels, with patients self-assessing readiness to progress.

The primary outcome is the change in the plyometric quotient, a measure of functional ability, based on a jump test using a force platform at 0 and 12 weeks. Secondary outcomes include dynamic strength, jump height, patient-reported symptoms (via questionnaires), return to sport, training compliance, adverse events, pain thresholds, re-injury rates, and psychological readiness for sports. Assessments will occur at baseline, 12 weeks, and 52 weeks.

DETAILED DESCRIPTION:
This trial is a randomised clinical trial with a 12-week intervention. The trial will be conducted at the Department of Physiotherapy, University College of Northern Denmark, Aalborg, Denmark. Participants will be stratified by their condition and block randomised (block sizes of 2 to 6) 1:1 to either 1) heavy-slow resistance training or 2) heavy-slow resistance training plus a plyometric exercise regimen. A researcher not involved in the trial will generate the allocation sequence using a random number generator and is the only person who will know the block sizes.

ELIGIBILITY:
Inclusion Criteria:

1. participants are required to perform either recreational running or participate in sports that include running or jumping activities (e.g., football, basketball, handball, volleyball) at least once per week for at least three months before inclusion
2. have had symptoms for at least three months
3. have pain/soreness with palpation of the tendon/fascia
4. mean pain during the past week of at least 2 on a 0 to 10 Numerical Rating Scale
5. pain during a pain provocation test (patellar tendinopathy: five single-legged decline squats, Achilles tendinopathy and plantar fasciopathy: ten single-legged heel raises)

Exclusion Criteria:

1. previous lower-extremity surgery
2. other lower-extremity musculoskeletal conditions that have required treatment by a healthcare professional during the past three months
3. pregnancy
4. diabetes
5. history of inflammatory systemic diseases (e.g., rheumatoid arthritis or spondylarthritis)
6. having received an injection with corticosteroid within the past six months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Plyometric quotient | From baseline to the 12-week follow-up
  The plyometric quotient is calculated by dividing the flight time by the contact time during single-leg hops and has good to excellent reliability. The test is performed on a force plate where the participant is instructed to perform 25 hops at a frequency of around two hops per second standing on their affected limb (or most symptomatic if they have bilateral symptoms). The first three and last two hops are excluded, which means that 20 hops are used to assess the flight time and contact time.

SECONDARY OUTCOMES:
Plyometric quotient | From baseline to the 52-week follow-up
  The plyometric quotient is calculated by dividing the flight time by the contact time during single-leg hops and has good to excellent reliability. The test is performed on a force plate where the participant is instructed to perform 25 hops at a frequency of around two hops per second standing on their affected limb (or most symptomatic if they have bilateral symptoms). The first three and last two hops are excluded, which means that 20 hops are used to assess the flight time and contact time.
Dynamic strength | Baseline to the 12-week and 52-week follow-ups
  Dynamic strength measured in knee extension and flexion and ankle plantar flexion by isokinetic dynamometry. The test is performed five times in each movement direction.
Drop countermovement jump height | From baseline to the 12-week and 52-week follow-ups
  Measured in centimetres and derived from the hop test (see description of the primary outcome) on the force plate.
Drop countermovement contact time | From baseline to the 12-week and 52-week follow-ups
  Measured in seconds and derived from the hop test (see description of the primary outcome) on the force plate.
Victorian Institute of Sports Assessment - Achilles (VISA-A) | Baseline to the 12-week and 52-week follow-ups
  Questionnaire only for participants with Achilles tendinopathy. Total score ranges from 0 to 100, where 100 indicates no pain or dysfunction and 0 represents severe limitations
TENDINS-A | From baseline to the 12-week and 52-week follow-ups
  Questionnaire only for participants with Achilles tendinopathy. The 13-item is scored between 0 and 100, with '0' representing a perfect score (no disability) and '100' representing complete disability.
Foot Health Status Questionnaire | Baseline to the 12-week and 52-week follow-ups
  Questionnaire only for participants with plantar fasciopathy. Includes four core domains: foot pain, foot function, footwear, and general foot health.
  Each domain is scored separately, ranging from 0 (poor foot health) to 100 (optimal foot health).
VISA-P | Baseline to the 12-week and 52-week follow-ups
  Questionnaire only for participants with patellar tendinopathy. Total score ranges from 0 to 100, with 100 indicating optimal function and 0 reflecting severe dysfunction.
Global Rating of Change | During the 12-week and 52-week follow-ups
  A 7-point numerical rating scale that evaluates participants' improvement compared to before treatment. Participants are dichotomised as improved if they rate themselves as 'much improved' or 'improved' (categories 6 and 7) and categorised as not improved if they rate themselves from 'slightly improved' to 'much worse' (categories 1 to 5)
Exercise compliance and fidelity | During the 12-week intervention.
  Based on training diaries. Exercise compliance relates to whether the training sessions have been performed, and fidelity relates to whether the exercises have been performed as prescribed regarding the number of repetitions, sets, and intensity.
Rate of return to sport | During the 12-week and 52-week follow-ups
  Measured by a self-developed questionnaire that includes questions regarding their physical performance and participation in sports
Adverse events | Throughout the time participants are enrolled (52 weeks)
  Adverse events will be collected throughout the trial and graded 1 to 5 according to the Common Terminology Criteria for Adverse Events v4.03. Participants are asked to contact the responsible clinician as soon as they experience any adverse event.
Pressure pain thresholds | From baseline to the 12-week and 52-week follow-ups
  Pressure pain thresholds measured by a pressure algometer on the tendon (Achilles or patella) or plantar fascia depending on the tendinopathy and the contralateral elbow. The test is performed with a handheld pressure algometer. The probe is placed perpendicular to the skin, and pressure is applied at a rate of 30 kPa/s. The participants are instructed to push the button of a hand-held switch when they first feel the sensation of pressure change to a sensation of pain, and the test is terminated
Re-injury | During the 12-week and 52-week follow-ups
  Rate of re-injury measured using the modified Oslo Sports Trauma Research Centre (OSTRC) Overuse Injury Questionnaire.
Psychological readiness to return to sport | Baseline to the 12-week and 52-week follow-ups
  Psychological readiness to return to sport measured by the Injury-Psychological Readiness to Return to Sport (I-PRRS) Scale. Participants respond to 10 items, depending on the version, related to confidence, emotional state, and readiness.
  Each item is scored on a scale of 0 to 100. 0 = Not confident/ready at all. 100 = Fully confident/ready

CONTACTS AND LOCATIONS:
Locations (1):
- University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon reasonable request.